CLINICAL TRIAL: NCT07357909
Title: A First-in-Human, Dose-Escalation Study to Evaluate the Safety and Tolerability of Intravenous Hydrogen-Oxygen Nanobubbles in Adults
Brief Title: Safety Study of Intravenous Hydrogen-Oxygen Nanobubbles in Adults
Acronym: NANO-SAFE
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Yayasan Inovasi Molekuler Indonesia (Indonesia Molecular Innovation Foundation) (Other)
Responsible Party: Principal Investigator, Olly Indrajani Dewi, Principal Investigator, Yayasan Inovasi Molekuler Indonesia (Indonesia Molecular Innovation Foundation)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: IMIF-202512-SiGNA-HHO-FIH
Record Dates: First submitted 2025-12-30; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Healthy Volunteer
Keywords: Hydrogen oxygen nanobubbles; Intravenous infusion; First-in-human study; Dose escalation; Safety; Tolerability; Healthy volunteers; Oxidative stress biomarkers; Tissue oxygenation; Redox biology

STUDY DESIGN:
Intervention Model Description: This is a sequential, dose-escalation study in which participants are enrolled in predefined cohorts. An initial sentinel cohort receives the lowest planned dose to confirm safety. Subsequent cohorts are enrolled sequentially and receive higher dose levels based on review of accumulated safety data from preceding cohorts. Dose escalation and cohort progression are guided by predefined safety review criteria. All participants receive the investigational intervention according to their assigned cohort, with structured safety monitoring following each administration.
Masking Description: This study is single-blind. Participants are blinded to the specific dose level of the investigational product they receive. Investigators and clinical staff are not blinded, as knowledge of the administered dose is required for safety monitoring, dose escalation decisions, and clinical management. No other parties are masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Intravenous Hydrogen-Oxygen Nanobubbles (Experimental): Participants in this single-arm study receive intravenous hydrogen-oxygen nanobubbles. The intervention is administered in two infusions given one week apart. Dose escalation is implemented across sequential cohorts based on review of accumulated safety data.
  Interventions: Other: Hydrogen-Oxygen Nanobubbles

INTERVENTIONS:
Other: Hydrogen-Oxygen Nanobubbles — Hydrogen-oxygen nanobubbles are administered as an intravenous infusion using standard clinical infusion equipment. Participants receive two infusions given one week apart according to the assigned dose cohort. Dose escalation across cohorts is guided by predefined safety review criteria.

SUMMARY:
The goal of this clinical trial is to learn whether hydrogen-oxygen nanobubbles can be safely given through a vein (intravenous infusion) to adults. This is a first-in-human study, meaning this type of infusion has not been tested in people before. The study focuses on safety and does not aim to treat or prevent any disease.

The main questions this study aims to answer are: 1) Can hydrogen-oxygen nanobubbles be given safely without causing serious or unacceptable side effects? 2) What dose range can be given safely to adults for future research?

About 40 adult participants, including healthy volunteers or people with mild, stable health conditions, will take part in the study. Each participant will receive two intravenous infusions, given one week apart. Some participants will receive a higher dose during the second infusion, depending on their assigned study group.

Researchers will closely monitor participants before, during, and after each infusion. This includes checking vital signs, heart activity, and blood tests. The study will also collect exploratory laboratory measurements, such as markers related to oxygen levels and oxidative stress, to help guide the design of future studies.

Participants will be followed for safety for about three weeks after starting the study. The information gained from this research will help determine whether hydrogen-oxygen nanobubbles can be studied further in clinical research.

DETAILED DESCRIPTION:
Hydrogen-oxygen nanobubbles (NB-HHO) are a novel gas-liquid formulation designed to deliver molecular hydrogen and oxygen in the form of nanoscale bubbles suspended in an aqueous solution. While molecular hydrogen administered by inhalation has been investigated in prior clinical and preclinical studies, the intravenous administration of hydrogen-oxygen nanobubbles has not previously been evaluated in humans. Preclinical investigations conducted by the study investigators in animal models have demonstrated the feasibility of intravenous NB-HHO administration and have not identified acute safety concerns at the dose ranges planned for initial human evaluation, supporting progression to a first-in-human clinical study.

This study is designed as a first-in-human, single-blind, dose-escalation clinical trial to characterize the safety, tolerability, and acceptable dose range of intravenously administered NB-HHO in adults. The study follows a predefined, safety-review-guided cohort progression strategy, with dose advancement contingent on review of accumulated safety data by a study safety review committee. The primary intent of this study is safety evaluation; it is not designed to assess clinical efficacy.

Participants will receive two intravenous administrations of NB-HHO, administered one week apart, according to the assigned dose cohort. A sentinel cohort is included to provide early safety confirmation at the lowest planned dose prior to enrollment of subsequent dose-escalation cohorts. Following the sentinel phase, sequential cohorts will evaluate higher second-dose levels while maintaining a consistent initial dose, allowing assessment of tolerability with within-participant dose escalation. This approach is intended to minimize risk while enabling efficient characterization of dose-related safety findings.

Intravenous infusions will be administered using standard clinical infusion equipment at a controlled infusion rate. Participants will undergo structured safety monitoring before, during, and after each infusion. Safety evaluations include clinical observation, vital sign measurements, electrocardiographic monitoring, and laboratory testing. Particular attention is given to infusion-related reactions, cardiopulmonary parameters, and laboratory indicators relevant to hematologic, hepatic, renal, coagulation, inflammatory, hemolytic, and complement activation pathways.

In addition to safety monitoring, the study incorporates exploratory physiological and biochemical assessments intended to characterize biological responses associated with NB-HHO administration. These exploratory evaluations include measurements related to tissue oxygenation, oxidative stress, and metabolic indicators. Data from these assessments are intended to support dose selection and inform the design of subsequent clinical studies; they are not intended to establish clinical efficacy.

Participant follow-up includes scheduled safety assessments after each infusion and continued observation following completion of dosing to identify any delayed or resolving adverse events. The overall study duration per participant is approximately three weeks from first infusion to completion of planned safety follow-up, with additional follow-up conducted as needed for unresolved safety findings.

The results of this study are expected to define a recommended dose range of NB-HHO suitable for further clinical investigation and to provide foundational human safety data to support future studies of this investigational platform.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 30 to 60 years at the time of enrollment.
* Judged to be healthy or to have mild, stable, well-controlled medical conditions based on medical history, physical examination, vital signs, and screening laboratory assessments.
* Body mass index (BMI) within 18.5 to 30.0 kg/m².
* Able and willing to comply with all study procedures and scheduled visits.
* Able to understand the study procedures and provide written informed consent prior to participation.

Exclusion Criteria:

* History or presence of clinically significant cardiovascular, pulmonary, neurological, hepatic, renal, hematologic, or immunologic disease that, in the investigator's judgment, could increase risk or interfere with study participation.
* Known history of stroke, transient ischemic attack, myocardial infarction, heart failure, or significant arrhythmia.
* Active infection, inflammatory condition, or febrile illness within 14 days prior to screening.
* Abnormal baseline laboratory findings considered clinically significant by the investigator.
* Known hypersensitivity or allergy to components of the investigational infusion or intravenous administration materials.
* Current or recent (within 30 days) participation in another interventional clinical study.
* Use of investigational drugs or therapies within 30 days prior to enrollment.
* Pregnancy or breastfeeding. Women of childbearing potential who are unwilling to use effective contraception during the study period.
* Any condition that, in the investigator's opinion, would make participation unsafe or compromise interpretation of study results.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Treatment-Emergent Adverse Events (TEAEs) | From first infusion (Day 0) through approximately 21 days after first infusion.
  Number and proportion of participants who experience one or more treatment-emergent adverse events following intravenous administration of hydrogen-oxygen nanobubbles. Adverse events will be assessed for severity, seriousness, and relationship to the investigational intervention.
Number of Participants With Clinically Significant Laboratory Abnormalities | From baseline through approximately 21 days after first infusion.
  Number of participants with laboratory test results that meet predefined criteria for clinically significant abnormalities following administration of hydrogen-oxygen nanobubbles. Laboratory assessments include hematology, renal function, hepatic function, coagulation parameters, markers of hemolysis, inflammatory markers, and complement activation markers.

SECONDARY OUTCOMES:
Change From Baseline in Oxidative Stress Biomarker: Malondialdehyde (MDA) | From baseline through approximately 21 days after first infusion.
  Change from baseline in blood malondialdehyde (MDA) concentration following intravenous administration of hydrogen-oxygen nanobubbles. MDA is used as a biomarker of lipid peroxidation and oxidative stress.
Change From Baseline in Antioxidant Enzyme Activity: Superoxide Dismutase (SOD) | From baseline through approximately 21 days after first infusion.
  Change from baseline in superoxide dismutase (SOD) activity measured in blood samples following administration of hydrogen-oxygen nanobubbles.
Change From Baseline in Nuclear Factor Erythroid 2-Related Factor 2 (Nrf2)-Related Biomarker Levels | From baseline through approximately 21 days after first infusion.
  Change from baseline in circulating Nrf2-related biomarker levels as an exploratory indicator of redox pathway activation following administration of hydrogen-oxygen nanobubbles.

CONTACTS AND LOCATIONS:
Locations (1):
- Ben Mari Hospital, Malang, East Java, Indonesia

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared publicly. De-identified data may be used for internal analyses and future research planning in accordance with applicable ethical approvals and data protection regulations.

REFERENCES:
- [Background] Hernowo, A. T., Widyarti, S., & Aristyani, S. (2024). Evaluating the safety and therapeutic efficacy of intravenous hydrogen nanobubble infusions in a hypercholesterolemic rat model. Berkala Penelitian Hayati, 30(1), 40-47.
- [Background] Aulanni'am, A., Riawan, W., Dyah Kinasih, W., Sri Widyarti, S., & Olly Indrayani, P. (2025). Uji Toksisitas Gelembung Nano Gasotransmitter. Institut Molekul Indonesia.
- [Background] Chan AW, Tetzlaff JM, Altman DG, Laupacis A, Gotzsche PC, Krleza-Jeric K, Hrobjartsson A, Mann H, Dickersin K, Berlin JA, Dore CJ, Parulekar WR, Summerskill WS, Groves T, Schulz KF, Sox HC, Rockhold FW, Rennie D, Moher D. SPIRIT 2013 statement: defining standard protocol items for clinical trials. Ann Intern Med. 2013 Feb 5;158(3):200-7. doi: 10.7326/0003-4819-158-3-201302050-00583. PMID 23295957
- [Background] Agustin V, Hernowo A. Stability evaluation of oxyhydrogen and hydrogen nanobubbles under thermal and pH stress conditions. Sci Rep. 2025 Dec 22;15(1):44273. doi: 10.1038/s41598-025-27868-z. PMID 41430413
- [Background] Food and Drug Administration, HHS. International Conference on Harmonisation; Guidance on M3(R2) Nonclinical Safety Studies for the Conduct of Human Clinical Trials and Marketing Authorization for Pharmaceuticals; availability. Notice. Fed Regist. 2010 Jan 21;75(13):3471-2. PMID 20349552
- [Background] Ohsawa I, Ishikawa M, Takahashi K, Watanabe M, Nishimaki K, Yamagata K, Katsura K, Katayama Y, Asoh S, Ohta S. Hydrogen acts as a therapeutic antioxidant by selectively reducing cytotoxic oxygen radicals. Nat Med. 2007 Jun;13(6):688-94. doi: 10.1038/nm1577. Epub 2007 May 7. PMID 17486089
- [Background] Ichihara M, Sobue S, Ito M, Ito M, Hirayama M, Ohno K. Beneficial biological effects and the underlying mechanisms of molecular hydrogen - comprehensive review of 321 original articles. Med Gas Res. 2015 Oct 19;5:12. doi: 10.1186/s13618-015-0035-1. eCollection 2015. PMID 26483953
- [Background] Agarwal A, Ng WJ, Liu Y. Principle and applications of microbubble and nanobubble technology for water treatment. Chemosphere. 2011 Aug;84(9):1175-80. doi: 10.1016/j.chemosphere.2011.05.054. PMID 21689840
- [Background] Szebeni J. Complement activation-related pseudoallergy caused by amphiphilic drug carriers: the role of lipoproteins. Curr Drug Deliv. 2005 Oct;2(4):443-9. doi: 10.2174/156720105774370212. PMID 16305447
- [Background] Szebeni J. Complement activation-related pseudoallergy: a new class of drug-induced acute immune toxicity. Toxicology. 2005 Dec 15;216(2-3):106-21. doi: 10.1016/j.tox.2005.07.023. Epub 2005 Sep 2. PMID 16140450
- [Background] Kensler TW, Wakabayashi N, Biswal S. Cell survival responses to environmental stresses via the Keap1-Nrf2-ARE pathway. Annu Rev Pharmacol Toxicol. 2007;47:89-116. doi: 10.1146/annurev.pharmtox.46.120604.141046. PMID 16968214
- [Background] Mattson MP. Hormesis defined. Ageing Res Rev. 2008 Jan;7(1):1-7. doi: 10.1016/j.arr.2007.08.007. Epub 2007 Dec 5. PMID 18162444
- [Background] Dragovic RA, Gardiner C, Brooks AS, Tannetta DS, Ferguson DJ, Hole P, Carr B, Redman CW, Harris AL, Dobson PJ, Harrison P, Sargent IL. Sizing and phenotyping of cellular vesicles using Nanoparticle Tracking Analysis. Nanomedicine. 2011 Dec;7(6):780-8. doi: 10.1016/j.nano.2011.04.003. Epub 2011 May 4. PMID 21601655